CLINICAL TRIAL: NCT03589092
Title: Genetic Causes of Gestational Diabetes in the Emirati Population
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Imperial College London Diabetes Centre (Other)
Responsible Party: Sponsor
Other Study IDs: IREC032
Record Dates: First submitted 2018-07-02; First posted 2018-07-17 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Gestational Diabetes; GDM; Maturity-onset Diabetes of the Young; MODY
Keywords: GDM; MODY; Genetic testing; Next Generation Sequencing; NGS
MeSH Terms: conditions — Diabetes, Gestational; Mason-Type Diabetes; Diabetes Mellitus, Type 2 | interventions — High-Throughput Nucleotide Sequencing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — DNA will be extracted from collected blood samples for genetic analysis

GROUPS / COHORTS (2):
- GDM Current: Currently pregnant women diagnosed with GDM.
  Next generation sequencing (NGS) methodologies will used on individuals suspected of genetic diabetes.
  Interventions: Genetic: Next generation sequencing (NGS)
- GDM History: Women with history of GDM (with negative GAD/IA2 antibodies if results available).
  Next generation sequencing (NGS) methodologies will used on individuals suspected of genetic diabetes.
  Interventions: Genetic: Next generation sequencing (NGS)

INTERVENTIONS:
Genetic: Next generation sequencing (NGS) — NGS Panel, Whole exome/genome sequencing

SUMMARY:
The study aims to identify the number of MODY patients to be found among Emirati women with GDM as the incidence and prevalence of monogenic diabetes among this group of patients is unknown. This will enable improvements in diagnostics, treatment and the counselling of these women.

DETAILED DESCRIPTION:
The present study aims to perform systematic genetic screening of genes known as the cause of MODY in women diagnosed with gestational diabetes to estimate the prevalence of MODY. This is important to understand the extent to which monogenic diabetes is encountered for the first time during pregnancy. Once women with MODY developing GDM have been identified, biomarkers to identify these women can be found which will assist the clinical process of performing genetic screening in the right subset of patients. Also for the women participating in the present study, this is of great importance as correct genetic diagnosis will provide them with the needed information to receive optimal treatment, correct plan for follow-up and a more accurate prognosis in relation to risk of future complication and therefore prevention of such.

ELIGIBILITY:
Inclusion Criteria:

* Currently pregnant women diagnosed with GDM.
* Women with history of GDM (with negative GAD/IA2 antibodies if results available).

Exclusion Criteria:

* Women with positive GAD/IA2 antibodies (if results available)
* Women genetically diagnosed as MODY

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women diagnosed with GDM, through Imperial College London Diabetes Centre (ICLDC) gestational diabetes clinic.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
GDM Identification | through study completion, an average of 2 year
  Identifying individuals with history of GDM or current diagnosis of GDM and analysing their GTT results and likelihood of MODY. GTT results will be extracted from patient's medical records.

SECONDARY OUTCOMES:
Next Generation Sequencing (NGS) | through study completion, an average of 2 year
  Next Generation Sequencing (NGS) technology will be applied to perform genetic testing, analysing 13 previously published MODY genes and potentially identifying novel causative mutations.
Novel diabetes genes | through study completion, an average of 2 year
  Identifying novel diabetes genes in the Emirati women with GDM by performing whole exome sequencing.
Genetic test results validation | through study completion, an average of 2 year
  Validating positive genetic test results by performing mutational analysis on parental, siblings and relatives samples. Request from parents, siblings and/or relatives to participate in the study will only occur if a novel (potentially pathogenic mutation) is identified and the primary participant agrees to it.
Potential biomarkers | through study completion, an average of 2 year
  Identifying potential biomarkers in women with MODY and who are developing GDM, to assist the selection of women suitable for genetic screening.
Prevalence of MODY | through study completion, an average of 2 year
  Determining the prevalence of MODY in women with GDM in the UAE.
Clinical outcomes determination | through study completion, an average of 2 year
  Determining the short and the long-term clinical outcomes of MODY in women with GDM in the UAE

CONTACTS AND LOCATIONS:
Overall Officials: Maha Barakat, PhD FRCP, Principal Investigator — Imperial College London Diabetes Centre; Torben Hansen, MD PhD, Principal Investigator — University of Copenhagen
Locations (1):
- Imperial College London Diabetes Centre, Abu Dhabi, United Arab Emirates